CLINICAL TRIAL: NCT01419743
Title: Randomized Controlled Trial: The Effects of Vitamin D Supplementation on In-vitro Fertilization Outcomes
Brief Title: Effect of Vitamin D Supplementation on In-vitro Fertilization (IVF) Outcomes
Status: Terminated | Type: Observational
Why Stopped: Low recruitment numbers
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Irene Moy, Clinical Fellow, Northwestern University
Other Study IDs: Moy 2011 Vit D
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Infertility; Vitamin D Deficiency
Keywords: Vitamin D deficiency; Supplementation; Infertility; Clinical pregnancy rates
MeSH Terms: conditions — Infertility; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- patients with Vit D level of < 20ng/mL: Group 1: randomized to receive 400 IU of vitamin D per day
- patients with Vit D levels <20ng/mL: Group 2: Randomized to receive 2000IU of Vitamin D per day
- patients with vit D levels between 20-30 ng/mL: Group 3: Randomized to receiving placebo
- patients with vit D levels between 20-30 ng/mL: Group 4: Randomized to receive 400IU of vitamin D per day
- patients with vit D levels between 20-30 ng/mL: Group 5: Randomized to receive 2000IU of vitamin D per day
- patients with vit D levels > 30ng/mL: Group 6: No treatment

SUMMARY:
Historically, vitamin D has been considered to play a role solely in bone and calcium metabolism. Numerous studies have suggested a link between vitamin D deficiency and adverse health outcomes such as malignancy, cardiovascular disease, immune functioning, and glucose metabolism. In the obstetrics literature, vitamin D deficiency has been linked to preeclampsia, gestational diabetes, and increased rate of cesarean section rate. Recent data from retrospective chart reviews have demonstrated a possible role of vitamin D in implantation and clinical pregnancy rates in patients undergoing in-vitro fertilization. Patients found to be deficient in vitamin D were found to have significantly lower clinical pregnancy rates when compared to patients who were replete in vitamin D levels. Currently, there are no prospective clinical trials investigating the effects of vitamin D supplementation on IVF outcomes such as clinical pregnancy rate and implantation rates. The investigators hypothesize that the vitamin D supplementation in patients found to be either deficient or insufficient in vitamin D will lead to improved pregnancy rates in infertility patients undergoing in-vitro fertilization.

DETAILED DESCRIPTION:
The trial will not pay for or subsidize for IVF treatment. Participants will receive blood Vitamin D screening test and any necessary supplements free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged ≤ 38 years undergoing fresh invitro fertilization cycles

Exclusion Criteria:

* Infertile women aged > 38 undergoing fresh invitro fertilization cycles
* Patients undergoing frozen embryo transfers
* Patients undergoing donor-egg cycles
* Patients who have a contraindication to receiving Vitamin D (e.g. patients with history of primary hyperparathyroidism, sarcoidosis, tuberculosis, kidney disease, or lymphoma)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women aged ≤ 38 years undergoing fresh in-vitro fertilization cycles
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | assessed at conclusion of the study (~ 1 yr)
  Serum hCG will be drawn per routine IVF protocol (~ 10 days after embryo transfer). Patients will have a repeat bHCG drawn 48hrs if they have a positive result from the first bHCG test. Clinical pregnancy will be defined as ultrasound documentation of fetal heart tones.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Kazer, MD, Principal Investigator — Northwestern Memorial Faculty Foundation; Irene Moy, MD, Study Chair — Northwestern University
Locations (3):
- United States (3):
  - Northwestern Memorial Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois

REFERENCES:
- [Background] Ozkan S, Jindal S, Greenseid K, Shu J, Zeitlian G, Hickmon C, Pal L. Replete vitamin D stores predict reproductive success following in vitro fertilization. Fertil Steril. 2010 Sep;94(4):1314-1319. doi: 10.1016/j.fertnstert.2009.05.019. Epub 2009 Jul 8. PMID 19589516
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Barrett H, McElduff A. Vitamin D and pregnancy: An old problem revisited. Best Pract Res Clin Endocrinol Metab. 2010 Aug;24(4):527-39. doi: 10.1016/j.beem.2010.05.010. PMID 20832734
- [Background] Heaney RP. Vitamin D in health and disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1535-41. doi: 10.2215/CJN.01160308. Epub 2008 Jun 4. PMID 18525006
- [Background] Johnson LE, DeLuca HF. Reproductive defects are corrected in vitamin d-deficient female rats fed a high calcium, phosphorus and lactose diet. J Nutr. 2002 Aug;132(8):2270-3. doi: 10.1093/jn/132.8.2270. PMID 12163674
- [Background] Kinuta K, Tanaka H, Moriwake T, Aya K, Kato S, Seino Y. Vitamin D is an important factor in estrogen biosynthesis of both female and male gonads. Endocrinology. 2000 Apr;141(4):1317-24. doi: 10.1210/endo.141.4.7403. PMID 10746634
- [Background] Halloran BP, DeLuca HF. Effect of vitamin D deficiency on fertility and reproductive capacity in the female rat. J Nutr. 1980 Aug;110(8):1573-80. doi: 10.1093/jn/110.8.1573. PMID 7400847
- [Background] Trivedi DP, Doll R, Khaw KT. Effect of four monthly oral vitamin D3 (cholecalciferol) supplementation on fractures and mortality in men and women living in the community: randomised double blind controlled trial. BMJ. 2003 Mar 1;326(7387):469. doi: 10.1136/bmj.326.7387.469. PMID 12609940
- [Background] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701
- [Background] Dobnig H, Pilz S, Scharnagl H, Renner W, Seelhorst U, Wellnitz B, Kinkeldei J, Boehm BO, Weihrauch G, Maerz W. Independent association of low serum 25-hydroxyvitamin d and 1,25-dihydroxyvitamin d levels with all-cause and cardiovascular mortality. Arch Intern Med. 2008 Jun 23;168(12):1340-9. doi: 10.1001/archinte.168.12.1340. PMID 18574092
- [Background] Bodnar LM, Catov JM, Simhan HN, Holick MF, Powers RW, Roberts JM. Maternal vitamin D deficiency increases the risk of preeclampsia. J Clin Endocrinol Metab. 2007 Sep;92(9):3517-22. doi: 10.1210/jc.2007-0718. Epub 2007 May 29. PMID 17535985